CLINICAL TRIAL: NCT02357784
Title: Sacral Neuromodulation in Dual Incontinence: Ultrasound and Afferent Nerve Sensation Assessment
Acronym: SaNDI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to low enrollment and the investigators want to explore a different primary objective
Sponsor: Northwestern University (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Principal Investigator, Margaret Mueller, Assistant Professor of Obstetrics and Gynecology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00098840
Record Dates: First submitted 2015-01-21; First posted 2015-02-06 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Dual Incontinence; Fecal Incontinence; Urinary Incontinence; Sacral Neuromodulation
Keywords: Sacral Neuromodulation; SNM; Dual Incontinence; Current Perception Threshold Testing; CPT Testing; Fecal Incontinence; Urinary Incontinence; Afferent Nerve Sensation; InterStim
MeSH Terms: conditions — Fecal Incontinence; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Current Perception Threshold Testing (Experimental): The subjects in this study will undergo Current Perception Threshold Testing and fill out several questionnaires both before their Sacral Nerve Modulator device implantation and again 3 months after the device implantation.
  Interventions: Device: Neurometer

INTERVENTIONS:
Device: Neurometer — The purpose of Current Perception Threshold (CPT) testing is to help physicians better understand how Sacral Neuromodulation affects the nerves of patients with dual incontinence. CPT Testing involves the use of a portable battery-operated machine which will stimulate the subject's nerves via an electrical stimulation. Electrodes will be placed via a catheter in to the subject's urethra and rectum, and the electrical current will be increased gradually until the subject feels the onset of tingling, buzzing, or warmth at the site of the electrode. The electrical current will then gradually decrease until no sensation of stimulation is felt. The procedure will then be repeated where the subject will be asked to hold the test button to increase the stimulus intensity above their sensory threshold (above the point where they can feel it) until the device automatically shuts off.
  Other Names: Neurometer CPT Testing; CPT Testing

SUMMARY:
Women with Dual Incontinence (DI) (both Urinary Incontinence (UI) and Fecal Incontinence (FI)) often have more bothersome symptoms, quality of life impact, and sexual dysfunction than those with just UI or FI. In many situations, DI is the result of a failure of communication between the brain and the sacral nerve, which controls the bladder, bowel, and pelvic floor. The only currently available treatment with level 1 effectiveness data for the treatment of BOTH UI and FI is called Sacral Neuromodulation (SNM). Sacral Neuromodulation is a standard of care treatment that involves surgically implanting a device in to a patient's body to target communication issues between their brain and bladder/bowel. Because the exact mechanism of action of SNM remains unclear, this study aims to better understand how SNM affects the nerves of patients with DI. Patients who are already planning on undergoing SNM device implantation will be recruited to this study. Study participants will undergo Current Perception Threshold (CPT) Testing and fill out questionnaires before SNM and 3 months after their SNM treatment. CPT Testing uses mild electrical stimulation in the urethra and rectum to measure and quantify the amount of physical stimuli required for the nerves in the pelvic floor to sense a stimulus. By learning more about nerve function in patients with DI, the investigators hope to find a way to screen patients before treatment with SNM to make sure the treatment will be effective for that individual.

DETAILED DESCRIPTION:
One in four women reports bothersome symptoms of a pelvic floor disorder with 16% reporting urinary incontinence (UI), otherwise known as leakage. Likewise, 1 in 5 women with UI reports fecal incontinence (FI). Women with dual incontinence (UI/FI) often have more bothersome symptoms, quality of life impact, and sexual dysfunction than those with just UI or FI. In many situations, bladder and/or bowel control problems are the result of a failure of communication between the brain and the sacral nerve. The sacral nerve controls the bladder, bowel, and pelvic floor and the muscles related to their function. If the brain and sacral nerve do not communicate correctly, the bladder and/or bowel cannot function properly, which often leads to incontinence, or leakage. The only currently available treatment with level 1 effectiveness data for the treatment of BOTH UI and FI is called Sacral Neuromodulation. Sacral Neuromodulation (SNM) is a standard of care procedure used to treat men and women that have symptoms of Urinary and Fecal Incontinence and involves surgically implanting a device in to the patient's body to target this communication problem by stimulating the nerves that control bladder and bowel function with mild electrical pulses. This helps the brain and nerves to communicate so the bladder and bowel can function properly. It is known that changes in nerve stimulation and muscular function are important factors in the cause and onset of UI and FI and in how a patient will respond to various treatments, however, the precise mechanism of action of SNM on UI and FI remains unclear.

This study therefore aims to obtain a better understanding of nerve and muscle function in patients with dual incontinence and to quantify how SNM affects the nerves of patients with dual incontinence. We hope to do so by using Current Perception Threshold (CPT) Testing, which is a way to quantify the function of different populations of afferent nerves. We will recruit patients who already plan on undergoing Sacral Neuromodulation implantation for the treatment of their dual incontinence, and as part of the research study we will use CPT testing to measure the amount of stimulation required to activate the participant's sacral nerve before SNM and will also measure the current perception threshold of the participant's sacral nerve after SNM treatment. We expect to see a difference in the amount of stimulation required to activate different pelvic floor nerves before and after the device implantation. By learning more about nerve function in patients with DI, we hope to find a way to screen patients before treatment with SNM to make sure the treatment will work for them. We also hope to learn how urethral and anal sphincter anatomy in patients with dual incontinence changes after treatment with SNM. Lastly, we will study the quality of sexual relationships in women with dual incontinence and their male partners and attempt to identify specific areas of dysfunction that are common in patients with DI.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female over the age of 18 years old
* Subject is diagnosed with idiopathic dual incontinence
* Subject is planning to undergo placement of a sacral nerve modulator
* Subject has at least 5 UUI episodes on a 3-day diary
* Subject has 2 FI episodes on a 7-day diary
* Subject has given signed, informed consent prior to registration on study

Exclusion Criteria:

* Subject has a neurologic disease
* Subject has a disease that may impair sphincter tone or sensation
* Subject is pregnant
* Subject has > Stage II pelvic organ prolapse
* Subject underwent rectal surgery in the past year
* Subject has chronic inflammatory bowel disease
* Subject has diathermy
* Subject has QTc prolongation
* Subject has cardiac arrhythmia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mueller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Group's Integrated Pelvic Health Program, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current Perception Threshold Testing
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Current Perception Threshold Testing
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urethral and Anal Afferent Nerve Innervation at 3 Months Post Sacral Neuromodulation Device Implantation
Time Frame: Baseline and 3 months Post-Treatment
Population: No data were collected
Arm/Group | Current Perception Threshold Testing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3-months
Description: There was only 1 arm of the study.
Arm/Group | Current Perception Threshold Testing
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT02357784/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02357784/SAP_001.pdf
  • Informed Consent Form (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT02357784/ICF_002.pdf